CLINICAL TRIAL: NCT06051942
Title: PRCT001 Aquablation theraPy Outcomes in pRostate Cancer patienTs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP0003
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostatic Hyperplasia; Localized Prostate Cancer
Keywords: AQUABEAM; AQUABEAM Robotic System; Aquablation; Aquablation therapy; Robotic Waterjet Treatment; RWT; Prostate cancer; Lower urinary tract symptoms; LUTS; BPH
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Aquablation (Experimental)
  Interventions: Device: Robotic Waterjet Treatment

INTERVENTIONS:
Device: Robotic Waterjet Treatment — The Aquablation therapy is a minimally invasive, image-guided, heat-free robotic therapy delivered by the AQUABEAM Robotic System. During Aquablation therapy, the AQUABEAM Handpiece is inserted transurethrally into the prostatic urethra. The operating physician then utilizes cystoscopy in conjunction with transrectal ultrasound (TRUS) imaging for real time visualization. The AQUABEAM Robotic System utilizes high-velocity sterile saline waterjet to resect and remove the prostate tissue according to the operating physician's treatment plan.
  Other Names: Aquablation therapy

SUMMARY:
The goal of this clinical trial is to assess the performance and safety of the AQUABEAM Robotic System for the resection and removal of prostate tissue in patients experiencing lower urinary tract symptoms (LUTS) and are diagnosed with localized prostate cancer. Participants will go through baseline and follow up assessments up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* International Prostate Symptom Score (IPSS) ≥ 8
* Gleason Grade Group 1-3
* Prostate-specific Antigen (PSA) ≤20ng/mL
* Cancer stage less than or equal to T2c

Exclusion Criteria:

* Patients with previous surgical treatment of benign prostatic hyperplasia
* MRI evidence of extracapsular extension of cancer
* Any severe illness that would prevent complete study participation or confound study results

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Clavien-Dindo Adverse Events (Percentage of Participants) Through 3 Months Post Treatment | 3 months post-treatment
  Proportion (percentage) of participants with adverse events rated as related to the study procedure classified as Clavien-Dindo Grade 2 or higher or any Grade 1 event resulting in persistent disability (ejaculatory disorder, erectile dysfunction, or incontinence) evidenced through 3 months post-treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - San Diego Clinical Trials, La Mesa, California
  - Endeavour Health (NorthShore University HealthSystem), Glenview, Illinois
  - Potomac Urology Center, Alexandria, Virginia
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- American University of Beirut, Beirut, Lebanon
- Tauranga Urology Research Ltd, Tauranga, New Zealand